CLINICAL TRIAL: NCT03567902
Title: A Randomized Trial on Comparison of Cervical Spine Motion During Tracheal Intubation Using Direct Laryngoscope Versus C-MAC Videolaryngoscope in Simulated Immobilized Cervical Spine
Brief Title: C-MAC Videolaryngoscope Intubation and Cervical Spine Motion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 1804-123-940
Record Dates: First submitted 2018-05-31; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Intubation;Difficult; Cervical Spinal Cord Injury
Keywords: C-MAC

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): C-MAC videolaryngoscope intubation -> Direct laryngoscope intubation
  Interventions: Device: C-MAC videolaryngoscope intubation; Device: Direct laryngoscope intubation
- Group B (Experimental): Direct laryngoscope intubation -> C-MAC videolaryngoscope intubation
  Interventions: Device: C-MAC videolaryngoscope intubation; Device: Direct laryngoscope intubation

INTERVENTIONS:
Device: C-MAC videolaryngoscope intubation — C-MAC videolaryngoscope intubation
Device: Direct laryngoscope intubation — Direct laryngoscope intubation

SUMMARY:
The aim of the study is to compare the effect of the C-MAC videolaryngoscope intubation technique vs. the conventional direct laryngoscope intubation technique on the cervical spine motion during intubation in patients with the simulated cervical immobilization.

DETAILED DESCRIPTION:
When the intubation is required in patients with an injured cervical spine, securing the airway while minimizing C-spine motion to prevent neurological damage can be very difficult. The awake intubation using a flexible bronchoscope is preferred as it minimizes C-spine motion. However, in the emergent clinical practice, direct laryngoscopy with manual in-line stabilization is most commonly used, because it is quicker and does not require patient collaboration. Numerous alternatives to direct laryngoscopy and fiberoptic bronchoscopy have been studied. But, none of these methods combines the convenience of direct laryngoscopy and the C-spine immobility afforded by intubation using a fiberoptic bronchoscope patient with an injured C-spine.

The videolaryngoscopy has recently developed extensively and become more widely available. It has the potential of combining the advantages of both direct laryngoscopy and intubation using a fiberoptic bronchoscope. Indeed, it provides an indirect view of the glottis, which could diminish C-spine movement, but its handling shares many similarities with direct laryngoscopy, which could make it more convenient than the flexible bronchoscope.

In the previous study examining C-spine movement during direct laryngoscopy and GlideScope® videolaryngoscopy, found no difference in movement at the rostral level but showed significantly less movement of the inferior C-spine with GlideScope® videolaryngoscopy. We postulate that C-MAC videolaryngoscope will induce less movement than direct laryngoscopy. The effect of C-MAC videolaryngoscope intubation technique on cervical spine motion is not investigated yet.

In this study, C-spine stabilization will be provided by Philadelphia neck collar. We will investigate a prospective cinefluoroscopic study comparing C-spine motion during direct laryngoscopy and C-MAC videolaryngoscope in patients with an intact C-spine stabilized by Philadelphia collar.

The duration and maximum change for C-MAC videolaryngoscope intubation technique was compared to those with direct laryngoscopy at each motion segment using a Student's paired t-test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists physical status of 1-2 and age of 20-80 years undergoing elective endovascular coiling to secure cerebral aneurysm under general anesthesia in neuroangiographic rooms.

Exclusion Criteria:

* Patients with C-spine injury, C-spine disease
* Patients with past medical history of C-spine surgery or intervention
* Patients with the upper airway abnormalities, such as inflammation, abscesses, tumours, polyps, or trauma.
* Patients with past medical history of gastro-oesophageal reflux disease and previous airway surgery, a high risk of aspiration, coagulation disorders, or Hunt Hess grade of 3-5.
* Body mass index > 30

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Maximum cervical spine motion (degree) | During tracheal intubation time, an expected average of 90 seconds
  Maximum angles measured at the occiput-C1, C1-C2, C2-C5 segments

SECONDARY OUTCOMES:
Intubation time | Within 90 seconds from insertion of device
  Check the intubation time (seconds) defines 'from insertion of device to oral cavity of patients to confirm successful intubation'
Number of intubation trial | During tracheal intubation time, an expected average of 1 minutes
  Check the number of intubation trial
Postoperative complications | During PACU stay time expected up to 1 hr
  Check the postoperative hoarseness, sore throat and numeric rating scale (1-10) we checked sore throat score
Postoperative complications | 24 hr after operation
  Check the postoperative hoarseness, sore throat and numeric rating scale (1-10) we checked sore throat score
Postoperative complications | After extubation, immediate postoperative period
  Blood tinged endotracheal tube ( yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: 82-2- 2072-2469 Park, Park, Principal Investigator — Seoul National University of Hospital

REFERENCES:
- [Background] Turkstra TP, Craen RA, Pelz DM, Gelb AW. Cervical spine motion: a fluoroscopic comparison during intubation with lighted stylet, GlideScope, and Macintosh laryngoscope. Anesth Analg. 2005 Sep;101(3):910-915. doi: 10.1213/01.ane.0000166975.38649.27. PMID 16116013
- [Background] Robitaille A, Williams SR, Tremblay MH, Guilbert F, Theriault M, Drolet P. Cervical spine motion during tracheal intubation with manual in-line stabilization: direct laryngoscopy versus GlideScope videolaryngoscopy. Anesth Analg. 2008 Mar;106(3):935-41, table of contents. doi: 10.1213/ane.0b013e318161769e. PMID 18292443
- [Background] Kim TK, Son JD, Seo H, Lee YS, Bae J, Park HP. A Randomized Crossover Study Comparing Cervical Spine Motion During Intubation Between Two Lightwand Intubation Techniques in Patients With Simulated Cervical Immobilization: Laryngoscope-Assisted Versus Conventional Lightwand Intubation. Anesth Analg. 2017 Aug;125(2):485-490. doi: 10.1213/ANE.0000000000001813. PMID 28244946
- [Derived] Paik H, Park HP. Randomized crossover trial comparing cervical spine motion during tracheal intubation with a Macintosh laryngoscope versus a C-MAC D-blade videolaryngoscope in a simulated immobilized cervical spine. BMC Anesthesiol. 2020 Aug 15;20(1):201. doi: 10.1186/s12871-020-01118-3. PMID 32799791